CLINICAL TRIAL: NCT01035307
Title: Genomic and Proteomic Profiling of Childhood AML
Brief Title: Studying Biomarkers in Tissue Samples From Young Patients With Acute Myeloid Leukemia Previously Enrolled on Clinical Trial POG-9421
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML09B2; COG-AAML09B2 (Other: Children's Oncology Group); CDR0000659560 (Other: NCI); NCI-2011-02201 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Collected for laboratory studies, including phospho-protein signaling and gene expression profiling studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genomic and Proteomic Profiling
  Interventions: Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: proteomic profiling; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in tissue samples from young patients with acute myeloid leukemia previously enrolled on clinical trial POG-9421.

DETAILED DESCRIPTION:
OBJECTIVES:

* To profile basal and potentiated phospho-protein networks (PPPNs) using tissue samples from pediatric patients with de novo acute myeloid leukemia (AML) previously enrolled on clinical trial POG-9421.
* To classify AML-based signal transduction mechanisms.
* To correlate profiles of basal and PPPNs with specific molecular lesions (e.g., FLT3-ITD, NPM, WT1, c-kit, CEPBα, PASGΔ75, and karyotype) and profiles of gene expression in tumor tissue samples.

OUTLINE: Banked tissue samples are collected for laboratory studies, including phospho-protein signaling and gene expression profiling studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia, meeting 1 of the following criteria:

  * Primary induction failure (i.e., failed to achieve remission within the first 60 days of therapy)
  * Relapsed disease (early or late)
  * In continuous complete remission
* Previously enrolled on POG-9421
* Tissue samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Previously enrolled on POG 9421
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Profiling of basal and potentiated phospho-protein networks (PPPNs) using tissue samples
Classification of AML-based signal transduction mechanisms
Correlation of basal and PPPN profiles with specific molecular lesions (e.g., FLT3-ITD, NPM, WT1, c-kit, CEPBα, PASGΔ75, and karyotype) and gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Norman J. Lacayo, MD, Principal Investigator — Stanford University